CLINICAL TRIAL: NCT01198418
Title: A Randomized Controlled Clinical Trial of an Internet-based Prevention Intervention to Reduce STI in High-risk HIV Infected MSM
Brief Title: A Web-based Intervention Study to Reduce High-risk Sexual Behavior by Persons Living With HIV AIDS (PLWH)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other); University of Southern California (Other); California HIV/AIDS Research Program (Other)
Responsible Party: Principal Investigator, Sheldon Morris, Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CCTG 592
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Sexually Transmitted Infections; HIV Infections
Keywords: STI; MSM; HIV; Prevention; Men having sex with men
MeSH Terms: conditions — Sexually Transmitted Diseases; HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Internet-based counseling (Experimental): Completes surveys monthly about their sexual and drug use behaviors as well as receives information designed to help reduce the chances of getting an STI.
  Interventions: Behavioral: Experimental
- Survey Alone (No Intervention): Completes surveys monthly about their sexual and drug use behaviors

INTERVENTIONS:
Behavioral: Experimental — Internet-based intervention that assesses transmission risk and provides prevention messages
  Arms: Internet-based counseling

SUMMARY:
This is a CCTG sponsored trial in collaboration with UCSD-AVRC investigators to get more information about the methods that are used on the internet to provide information on how to reduce the risk of giving or getting infections that are often or usually passed from one person to another during sexual or intimate contact (sexually transmitted infection (STI)). STIs include chlamydia, gonorrhea and syphilis. The purpose of this study is to develop methods that will allow someone who is living with HIV an easy way that they can get information and learn of ways on their own that can decrease their chances of getting sexually transmitted infections and ways that they can reduce the chance that they may transmit HIV to others.

DETAILED DESCRIPTION:
Design: CCTG 592 is a randomized, controlled study that will compare the efficacy of web-based intervention to reduce high-risk sexual behavior by persons living with HIV AIDS (PLWH).

Duration: 48 weeks

Sample Size: 200 subjects (100 per arm) that will be randomized

Study Population: HIV-1-infected men who have sex with men (MSM) at least 18 years of age who have a recent history of transmission risk behavior.

Stratification: Subjects will be stratified based upon their baseline antiretroviral use, whether they have a home computer and by site.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection, as documented by any licensed screening antibody test, such as ELISA, and confirmed by a second antibody test, such as Western blot, or detectable plasma HIV-1 RNA at any time prior to study entry. If an ELISA or Western Blot are not available, HIV infection may be documented by two HIV RNA values > 2000 copies/mL, drawn at least 24 hours apart. The HIV RNA assays should have been run at a CLIA approved laboratory or equivalent.
* 18 years of age or older.
* Male.
* At least one of the following:
* An HIV negative or unknown status sexual partner in the past three months.
* A sexually transmitted disease in the past 1 year (other than HIV).
* More than 2 male partners in past year.
* Unprotected anal sex in past 3 month.
* Capable of signing written informed consent.
* Read and comprehend English
* Adequate computer skills for study.

Exclusion Criteria:

* Uncontrolled psychiatric condition.
* Drug or alcohol users with use that in the opinion of the investigator, would limit follow-up and adequate consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2010-07-09 (Actual); Primary Completion 2017-10-18 (Actual); Study Completion 2017-11-09 (Actual)

PRIMARY OUTCOMES:
STI incidence | Baseline and follow-up visits every 3 months
  * To compare the composite STI incidence of syphilis or Chlamydia trachomatis (CT) or Neisseria gonorrhea (GC) at any mucosal site among sexually active HIV-infected men during 12 months participation in an Internet risk reduction intervention compared to those that receive a survey instrument alone.
  * To compare the incidence of nonspecific urethritis by urinalysis and testing for Mycoplasma genitalum and trichomonas sp. among sexually active HIV-infected men during 12 months participation in an Internet risk reduction intervention compared to those that receive a survey instrument alone.

SECONDARY OUTCOMES:
Evaluate risk factors of STIs | Baseline, follow-up visits every 3 months
  * Compare:a)self reported levels of unsafe sex among HIV-infected men b)intention to start ARV among HIV-infected men not currently on ARV will increase during 12 mos. participation in an internet risk reduction intervention compared to survey instrument alone
  * Compare self-reported among HIV-infected men during 12 mos. participation as measured by those reporting 100% disclosure in an internet risk reduction intervention compared to survey instrument alone
  * Collect genital tract secretions of semen for future study

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Morris, MD, MPh, Principal Investigator — UC San Diego AntiViral Research Center (AVRC); Joel Milam, PhD, Study Chair — University of California, San Diego
Locations (3):
- United States (3):
  - University of Southern California, Los Angeles, California
  - University of California, San Diego, San Diego, California
  - University of California, Los Angeles (Harbor), Torrance, California

REFERENCES:
- See also: (organization's website) — https://www.cctg.ucsd.edu